CLINICAL TRIAL: NCT00878878
Title: A Phase 4, Placebo Controlled, Single-blind, Cross-over Safety Study to Evaluate the Effect of Optison on Pulmonary Artery Systolic Pressure (PASP) and Pulmonary Vascular Resistance (PVR) as Measured by Right Heart Catheterization
Brief Title: Evaluate Effect of Optison on Pulmonary Artery Systolic Pressure (PASP) and Pulmonary Vascular Resistance (PVR).
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GE Healthcare (Industry)
Collaborators: ICON Clinical Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: GE-191-004
Record Dates: First submitted 2009-04-08; First posted 2009-04-09 (Estimated); Results first posted 2012-08-24 (Estimated); Last update posted 2012-08-24 (Estimated); Status verified 2012-07

CONDITIONS: Pulmonary Hypertension
Keywords: Pulmonary artery systolic pressure (PASP); Pulmonary Vascular Resistance (PVR); Right Heart Catheterization; Pulmonary hemodynamics
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — FS 069; Glucose

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Experimental)
  Interventions: Drug: Optison (Perflutren Protein-Type A Microspheres Injectable Suspension); Drug: Dextrose
- Arm B (Experimental)
  Interventions: Drug: Optison (Perflutren Protein-Type A Microspheres Injectable Suspension); Drug: Dextrose

INTERVENTIONS:
Drug: Optison (Perflutren Protein-Type A Microspheres Injectable Suspension) — Arm A: Single intravenous (IV) injection of 0.5 mL Optison followed by single IV injection of 0.5 mL 5% dextrose.
  Arm B: Single IV injection of 0.5 mL 5% dextrose followed by single IV injection of 0.5 mL Optison.
  Other Names: Perflutren Protein-Type A Microspheres Injectable Suspension
Drug: Dextrose — Arm A: Single intravenous (IV) injection of 0.5 mL Optison followed by single IV injection of 0.5 mL 5% dextrose.
  Arm B: Single IV injection of 0.5 mL 5% dextrose followed by single IV injection of 0.5 mL Optison.

SUMMARY:
The design of this study is to conduct a comprehensive safety evaluation of the pulmonary hemodynamic effects of Optison. The study is being conducted in subjects referred for cardiac catheterization for clinical reasons.

ELIGIBILITY:
Inclusion Criteria:

* Must be already scheduled for left and/or right heart catheterization for clinical reasons.
* Must be in sinus rhythm, without an arrhythmia likely to affect the ability to assess pulmonary hemodynamics by catheterization, as determined by the investigator.
* Women of childbearing potential must be using adequate birth control and have a negative pregnancy test.

Exclusion Criteria:

* History of right-to-left, bi-directional, or transient right-to-left cardiac shunts or diagnosed by color flow Doppler echocardiography during screening.
* Hypersensitivity to Optison, perflutren, blood, blood products, or albumin.
* Female subjects who are nursing mothers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-03; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Jefferds, Study Director — ICON Development Solutions
Locations (1):
- ICON Development Solutions, Elliott, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Optison First, Then Followed by Placebo Control: Optison product (Perflutren Protein-Type A Microspheres Injectable Suspension, USP) given first, than the Placebo Control (5% Dextrose). There was a 15 minute interval between the injections.
- Placebo Control First, Then Followed by Optison Product: Placebo Control (5% Dextrose) was used first, then the Optison product (Perflutren Protein-Type A Microspheres Injectable Suspension, USP). There was a 15 minute interval between the injections.
Period: Overall Study
Arm/Group | Optison First, Then Followed by Placebo Control | Placebo Control First, Then Followed by Optison Product
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Optison First, Then Followed by Placebo Control | Placebo Control First, Then Followed by Optison Product | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 8 | 17
  >=65 years | 6 | 7 | 13
Age Continuous [Mean (Standard Deviation); unit: years] | 53 (16.1) | 60 (16.7) | 57 (16.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 16
  Male | 8 | 6 | 14
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Observed the Change of Pulmonary Artery Systolic Pressure (PASP) Measured by Millimeters of Mercury (mm hg) Within Certain Time Periods. This is Per Sequence and Not a Cross-over Study.
Description: Measurement of the Pulmonary artery systolic pressure (PASP) results, which were taken from the subject in millimeters of mercury; a unit of pressure (mm hg), at Baseline and at 2 minutes, 6 minutes and 10 minutes. This is per sequence and not a cross-over study.
Time Frame: Measurements recorded at Baseline, 2 minutes, 6 minutes and 10 minutes post contrast administration
Population: The Pulmonary artery systolic pressure (PASP) results were taken at Baseline and at 2 minutes, 6 minutes and 10 minutes.
Measure: Mean (Standard Deviation); unit: mm Hg
Groups:
- Optison Given First, Then Placebo Control (5%Dextrose): Optison product (Perflutren Protein-Type A Microspheres Injectable Suspension, USP) was given first followed by the Placebo Control (5% Dextrose). There was a 15 minute interval between the injections.
- Placebo Control (5% Dextrose) Given First, Then Optison: Placebo Control (5% Dextrose) was given first followed by the Optison product (Perflutren Protein-Type A Microspheres Injectable Suspension, USP). There was a 15 minute interval between the injections.
Arm/Group | Optison Given First, Then Placebo Control (5%Dextrose) | Placebo Control (5% Dextrose) Given First, Then Optison
Number analyzed (Participants) | 15 | 15
mm Hg
  PASP (Units: mmHg) - Baseline | 55.2 (28.1) | 53.7 (27.1)
  2 min Post | 55.6 (27.9) | 53.8 (26.9)
  6 min Post | 54.1 (28.1) | 54.6 (27.7)
  10 min Post | 54.57 (27.0) | 54.9 (27.6)

2. Secondary Outcome: Recorded Any Adverse Events From the Optison and Control Solution (5% Dextrose) Used in Subjects With Normal and Elevated Pulmonary Artery Systolic Pressure (PASP. This is Per Sequence and Not a Cross-over Study.
Description: Observe subjects with normal pulmonary artery systolic pressure (PASP) and elevated pulmonary artery systolic pressure (PASP) as measured by any adverse events.
  The number of participants were stratified based on a screening pulmonary artery systolic pressure (PASP). Subjects stratified by; 11 subjects that were Normal PASP and 19 subjects that were Elevated PASP.
  This is per sequence and not a cross-over study.
Time Frame: During the injection and catheterization procedure, and for up to 24 hours post-injection
Population: The number of participants were stratified based on a screening pulmonary artery systolic pressure (PASP). Subjects stratified by; Normal PASP and Elevated PASP.
Measure: Number; unit: Adverse Events
Groups:
- Normal Pulmonary Artery Systolic Pressure (PASP): Observe subjects with normal pulmonary artery systolic pressure (PASP)as measured by any adverse events. The number of participants were stratified based on a screening pulmonary artery systolic pressure (PASP).
- Elevated Pulmonary Artery Systolic Pressure (PASP): Observe subjects with elevated pulmonary artery systolic pressure (PASP)as measured by any adverse events. The number of participants were stratified based on a screening pulmonary artery systolic pressure (PASP).
Arm/Group | Normal Pulmonary Artery Systolic Pressure (PASP) | Elevated Pulmonary Artery Systolic Pressure (PASP)
Number analyzed (Participants) | 11 | 19
Adverse Events
  Subjects with Serious adverse event up to 24h post | 0 | 0
  Subjects with adverse event-up to 24h post | 0 | 1

3. Primary Outcome: Observed the Change of Pulmonary Vascular Resistance (PVR) Measured by Wood Units Within Certain Time Periods. This is Per Sequence and Not a Cross-over Study.
Description: Measurement of the pulmonary vascular resistance (PVR) results, which was taken from the subject in Wood Units, taken at Baseline and at 2 minutes, 6 minutes and 10 minutes. This is per sequence and not a cross-over study.
Time Frame: Measurements recorded at Baseline, 2 minutes, 6 minutes and 10 minutes post contrast administration
Population: The pulmonary vascular resistance (PVR) results were taken at Baseline and at 2 minutes, 6 minutes and 10 minutes.
Measure: Mean (Standard Deviation); unit: Wood Units
Arm/Group | Optison Given First, Then Placebo Control (5%Dextrose) | Placebo Control (5% Dextrose) Given First, Then Optison
Number analyzed (Participants) | 15 | 15
Wood Units
  PVR (Units: Wood Units) - Baseline | 3.6 (2.9) | 3.9 (4.0)
  2 min Post | 3.67 (3.56) | 3.9 (4.4)
  6 min Post | 3.3 (2.9) | 3.87 (3.68)
  10 min Post | 3.8 (3.4) | 3.5 (3.3)

ADVERSE EVENTS:
Groups:
- Optison Product First Followed by Placebo Control (5%Dextrose): Optison product (Perflutren Protein-Type A Microspheres Injectable Suspension, USP) given first followed by the Placebo Control (5% Dextrose). There was a 15 minute interval between the injections.
- Placebo Control (5% Dextrose) First Followed by the Optison: Placebo Control (5% Dextrose) given first followed by the Optison product (Perflutren Protein-Type A Microspheres Injectable Suspension, USP. There was a 15 minute interval between the injections.
Arm/Group | Optison Product First Followed by Placebo Control (5%Dextrose) | Placebo Control (5% Dextrose) First Followed by the Optison
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 1/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Optison Product First Followed by Placebo Control (5%Dextrose) (N=15) | Placebo Control (5% Dextrose) First Followed by the Optison (N=15)
Procedural Pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No